CLINICAL TRIAL: NCT05638230
Title: Relative Importance of Cardiovascular Risk Factors and Echocardiographic Parameters Affecting Left Atrial Strain
Acronym: RICH-LAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Minkwan Kim, MD, Clinical assistant professor, Yonsei University
Other Study IDs: 9-2022-0101
Record Dates: First submitted 2022-10-24; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure, Diastolic; Heart Failure, Preserved Ejection Fraction
Keywords: left atrial reservoir strain; HFA-PEFF; LA strain; Heart failure with preserved ejection fraction (HFpEF)
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIgh HFA-PEFF points (≥5)
  Interventions: Diagnostic Test: Left atrial reservoir strain
- Low to intermediate HFA-PEFF points (<5)
  Interventions: Diagnostic Test: Left atrial reservoir strain

INTERVENTIONS:
Diagnostic Test: Left atrial reservoir strain — LA strain measurements can be obtained by two dimensional (2D) speckle tracking echocardiography (STE). Longitudinal strain and strain rate curves are generated for each of six atrial segments, obtained from the apical four and two chamber views.
  In the reservoir phase, as the LA fills and stretches, there is positive atrial strain that reaches its peak in systole at the end of LA filling, prior to opening of the mitral valve. Following this, passive LA emptying ensues with opening of the mitral valve resulting in decreased atrial strain with negative deflection of the strain curve up to a plateau period which is analogous to diastasis. LA reservoir strain (LARS), or peak atrial longitudinal strain or LA systolic strain, is measured at the end of the reservoir phase.

SUMMARY:
The goal of this observational study is to learn about left atrial reservoir strain in patients with heart failure with preserved ejection fraction. The main questions it aims to answer are:

* Usefullness of LARS as a predictor of high HFA-PEFF diagnostic algorithm scores (≥5)
* The relative importance of LARS in variables including each component of HFA-PEFF and traditional cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ICD-10 code of heart failure (I50) from August 2021 to July 2022
* 20-year-old or higher age
* Participants who are available to measure left atrial reservoir strain

Exclusion Criteria:

* Left ventricular ejection fraction <50%
* Supraventricular arrhythmia (e.g. atrial flutter/fibrillation, atrial tachycardia)
* Participants who are given pacemaker or ICD implantation procedure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited a cardiovascular center clinic for dyspnea and chest discomfort and who underwent echocardiography were enrolled for participants suspected of having heart failure with preserved ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Statistical significant of LA reservoir strain to estimate high HFA-PEFF score (≥5) | through study completion, an average of 1 year
  Statistical significant of LA reservoir strain to estimate high HFA-PEFF score (≥5) in multiple linear regression analysis.
Relative importance of left atrial reservoir strain | through study completion, an average of 1 year
  Relative importance of left atrial reservoir strain among variables, including component of HFA-PEFF score, using supervised machine learning algorithm (random forest analysis) to estimate high HFA-PEFF score (≥5). LA reserver strain was measured using Automated Functional Imaging (AFI) of the left atrium 3.0 version (GE Healthcare)

CONTACTS AND LOCATIONS:
Locations (1):
- Minkwan Kim, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim M, Bae S, Park JH, Jung IH. Relative importance of left atrial reservoir strain compared with components of the HFA-PEFF score: a cross-sectional study. Front Cardiovasc Med. 2023 Oct 12;10:1213557. doi: 10.3389/fcvm.2023.1213557. eCollection 2023. PMID 37900564